CLINICAL TRIAL: NCT00319748
Title: Phase II Study of 852A Administered Subcutaneously in Patients With Metastatic Refractory Breast, Ovarian, Endometrial and Cervical Cancers
Brief Title: Study of Immune Response Modifier in the Treatment of Breast, Ovarian, Endometrial and Cervical Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Melissa Geller, M.D., Masonic Cancer Center, University of Minnesota
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06US03IMP-852A; MT2006-02 (Other: Blood and Bone Marrow Transplantation Program); 2006LS005 (Other: Masonic Cancer Center, University of Minnesota); NCT00363493 (obsolete NCT alias)
Record Dates: First submitted 2006-04-27; First posted 2006-04-27 (Estimated); Results first posted 2009-09-25 (Estimated); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Breast Cancer; Ovarian Cancer; Endometrial Cancer; Cervical Cancer
Keywords: Breast; Ovarian; Endometrial; Cervical; Metastatic; 852A; IRM; Oncology; Metastatic Cervical Cancer; Metastatic Ovarian Cancer; Metastatic Breast Cancer; Metastatic Endometrial Cancer
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Endometrial Neoplasms; Uterine Cervical Neoplasms; Neoplasm Metastasis; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intent-To-Treat (Experimental): Patients treated with at least one dose - 852A subcutaneous injection.
  Interventions: Drug: 852A
- Evaluable Cohort (Experimental): Patients who received all 24 doses of 852A per protocol.
  Interventions: Drug: 852A

INTERVENTIONS:
Drug: 852A — 0.2% 852a subcutaneous injection, 2 times per week for 12 weeks (24 doses) starting at 0.6 mg/m2; subsequent dose escalation for additional courses may be increased by 0.2 mg/m2 not to exceed 1.2 mg/m2.
  Other Names: TLR-7; Toll-like receptor-7

SUMMARY:
The purpose of this study is to evaluate the anti-tumor activity of 852A when used to treat metastatic breast, ovarian, endometrial or cervical cancer not responding to standard treatment.

DETAILED DESCRIPTION:
852A will be administered as a subcutaneous injection (SC) 2 times per week for 12 weeks (24 doses) with provisions for dose escalation or reduction based on tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Adequate performance status:

  * Breast - Karnofsky score > 50;
  * Ovarian, endometrial or cervical - Gynecologic Oncology Group (GOG) performance score ≤2
* If female and of childbearing potential, are willing to use adequate contraception (hormonal, barrier method, abstinence) prior to study entry and for the duration of study participation.
* Normal organ function within 14 days of study entry
* Diagnosis of one of the following malignancies:

  * Metastatic breast cancer (BR)
  * Metastatic ovarian cancer (OV)
  * Metastatic endometrial cancer (EM)
  * Metastatic cervical cancer (CX)

Breast Cancer Inclusion Criteria:

* Measurable metastatic disease (>1cm) in at least one site other than bone-only
* Progression on or failure to respond to at least one previous chemotherapy regimen for metastatic disease
* Progression on prior therapy with a hormonal agent if estrogen receptor or progesterone receptor positive, and/or with trastuzumab if HER2-neu positive. If patient has progressed through hormone or trastuzumab therapy only, must have received one chemotherapy regimen.

Ovarian Cancer Inclusion Criteria:

* Measurable metastatic disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST)
* Primary tumor must have been diagnosed histologically as either epithelial ovarian cancer, fallopian tube cancer, or primary peritoneal cancer (not borderline or low malignant potential epithelial carcinoma).
* Subjects must have failed at least two previous chemotherapy regimens. Paclitaxel must have been a component of one or both regimens and cisplatin or carboplatin must have been a component of one or both regimens.

Endometrial Cancer Inclusion Criteria:

* Measurable metastatic disease
* Histologically proven recurrent or persistent endometrial cancer that is not amenable to curative treatment with surgery and/or radiation therapy AND has failed 2 previous treatment regimens

Cervical Cancer Inclusion Criteria:

* Measurable metastatic disease
* Histologically proven recurrent or persistent squamous cell carcinoma, adenosquamous carcinoma, or adenocarcinoma of the cervix that is not amenable to curative treatment with surgery and/or radiation therapy AND has failed 2 previous treatment regimens.

Exclusion Criteria:

* Had/have the following prior/concurrent therapy:

  * Systemic corticosteroids (oral or injectable) within 7 days of first dose of 852A (topical or inhaled steroids are allowed)
  * Investigational drugs/agents within 14 days of first dose of 852A
  * Immunosuppressive therapy, including cytotoxic agents within 14 days of first dose of 852A (nitrosoureas within 30 days of first dose)
  * Drugs known to induce QT interval prolongation and/or induce Torsades de pointes unless best available drug required to treat life-threatening conditions
  * Radiotherapy within 3 weeks of the first dose of 852A
  * Hematopoietic cell transplantation within 4 weeks of first dose of 852A
  * Evidence of active infection within 3 days of first dose of 852A
  * Active fungal infection or pulmonary infiltrates (prior treated disease stable for 2 weeks is allowable)
  * Cardiac ischemia, cardiac arrhythmias or congestive heart failure uncontrolled by medication
  * History of, or clinical evidence of, a condition which, in the opinion of the investigator, could confound the results of the study or put the subject at undue risk
  * Uncontrolled intercurrent or chronic illness
  * Active autoimmune disease requiring immunosuppressive therapy within 30 days
  * Active coagulation disorder not controlled with medication
  * Pregnant or lactating
  * Concurrent malignancy (if in remission, at least 5 years disease free) except for localized (in-situ) disease, basal carcinomas and cutaneous squamous cell carcinomas that have been adequately treated
  * Any history of brain metastases or any other active central nervous system (CNS) disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2006-04; Primary Completion 2007-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Cooley, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota; Melissa A. Geller, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 15 patients were originally consented to enter the study; however 1 patient died before participating in study and 1 patient made the decision to withdraw before being treated.
Groups:
- Patients Treated With 852A: Patients that received at least one dose of study treatment with 852A (0.6 mg/m^2 to 1.2 mg/m^2 dose, 2 times/week for 12 weeks).
Period: Overall Study
Arm/Group | Patients Treated With 852A
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Patients Treated With 852A Study Drug: Patients that received at least one dose of study treatment with 852A (0.6 mg/m^2 to 1.2 mg/m^2 dose, 2 times/week for 12 weeks).
Arm/Group | Patients Treated With 852A Study Drug
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 52 (9.6) [24 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Patients With Tumor Response (Response Evaluation Criteria in Solid Tumors) Who Received All 24 Doses of 852A.
Description: Assessment of anti-tumor activity of 852A using Response Evaluation Criteria in Solid Tumors (RECIST) criteria to evaluate tumor response after 24 doses. Complete Response (CR)= disappearance of all target lesions, Partial Response (PR) = at least 30% decrease in sum of longest diameter of target lesions, Progressive Disease (PD) = at least 25% increase in sum of longest diameter of target lesions, Stable Disease = neither PR or PD.
Time Frame: after 12 weeks (24 doses of 852A)
Population: Includes only patients that received all 24 doses of 852A.
Measure: Number; unit: Participants
Groups:
- Patients With Ovarian Cancer: Participants with ovarian cancer who received all 24 doses of 852A.
Arm/Group | Patients With Ovarian Cancer
Number analyzed (Participants) | 3
Participants
  Complete Response | 0
  Partial Response | 0
  Stable Disease | 1
  Progressive Disease | 2

2. Secondary Outcome: Mean Difference Values for Interleukin 1 Receptor Antagonist (IKL1ra)
Description: Measures the difference of IL1ra (cytokine) values as a means of immune activation pre-treatment and 6 hours post-treatment in patients that received at least one dose of study treatment with 852A.
Time Frame: Prior to Dose 1 and 6 hours after Dose 1
Population: One patient did not have value reported at 6 hours after treatment, so cannot be included.
Measure: Mean (95% Confidence Interval); unit: pg/mL
Groups:
- Patients Treated With 852A: Difference in range values from pre-treatment to post-treatment for cytokine level of IL1ra in patients treated with 852A.
Arm/Group | Patients Treated With 852A
Number analyzed (Participants) | 12
pg/mL | 6265.10 [-1105.01 to 13635.21]

3. Secondary Outcome: Mean Difference Values for 10 kDa Interferon-gamma-induced Protein (IP-10)
Description: Measures differences in IP-10 (cytokine) values as a means of immune activation pre-treatment and 6 hours post-treatment in patients that received at least one dose of study treatment with 852A.
Time Frame: Prior to Dose 1 and 6 Hours Post-Dose
Population: One patient did not have a value reported at 6 hours after treatment so cannot be included in analysis.
Measure: Mean (95% Confidence Interval); unit: pg/mL
Groups:
- Patients Treated With 852A: Difference in range values from pre-treatment to post-treatment for cytokine level of IP-10 in patients treated with 852A.
Arm/Group | Patients Treated With 852A
Number analyzed (Participants) | 12
pg/mL | 1685.96 [546.82 to 2825.10]

4. Secondary Outcome: Mean Difference Values for Macrophage Inflammatory Protein-1 Alpha (MIP-1a)
Description: Measures difference in MIP-1a (cytokine) values as a means of immune activation pre-treatment and 6 hours post-treatment in patients that received at least one dose of study treatment with 852A.
Time Frame: Prior to Dose 1 and 6 Hours Post-Dose
Population: Only 5 patients had a value reported at 6 hours after treatment.
Measure: Mean (95% Confidence Interval); unit: pg/mL
Groups:
- Patients Treated With 852A: Difference in range values from pre-treatment to post-treatment for Macrophage Inflammatory Protein-1 Alpha (cytokine) level in patients treated with 852A.
Arm/Group | Patients Treated With 852A
Number analyzed (Participants) | 5
pg/mL | 95.72 [-50.77 to 242.20]

5. Secondary Outcome: Mean Difference Values for Macrophage Inflammatory Protein-1 Beta (MIP-1b)
Description: Measures difference in Macrophage Inflammatory Protein-1 Beta (cytokine) values as a means of immune activation pre-treatment and 6 hours post-treatment in patients that received at least one dose of study treatment with 852A.
Time Frame: Prior to Dose 1 and 6 Hours Post-Dose
Population: Two patients did not have recorded values at 6 hours after treatment so cannot be included in analysis.
Measure: Mean (95% Confidence Interval); unit: pg/mL
Groups:
- Patients Treated With 852A: Difference in range values from pre-treatment to post-treatment for cytokine level of MIP-1b in patients treated with 852A.
Arm/Group | Patients Treated With 852A
Number analyzed (Participants) | 11
pg/mL | 141.04 [-95.72 to 377.84]

6. Secondary Outcome: Mean Difference Values for Soluble CD40 Ligand (sCD40L)
Description: Measures difference in Soluble CD40 ligand (cytokine) values as a means of immune activation pre-treatment and 6 hours post-treatment in patients that received at least one dose of study treatment with 852A.
Time Frame: Prior to Dose 1 and 6 Hours Post-Dose
Population: One patient did not have recorded value at 6 hours after treatment and cannot be included in analysis.
Measure: Mean (95% Confidence Interval); unit: pg/mL
Groups:
- Patients Treated With 852A: Difference in range values from pre-treatment to post-treatment for cytokine level of sCD40L in patients treated with 852A.
Arm/Group | Patients Treated With 852A
Number analyzed (Participants) | 12
pg/mL | -1061.96 [-5110.99 to 29878.08]

7. Secondary Outcome: Mean Difference Values for Tumor Necrosis Factor-alpha (TNF-a)
Description: Measures difference in Tumor necrosis factor-alpha (cytokine) values as a means of immune activation pre-treatment and 6 hours post-treatment in patients that received at least one dose of study treatment with 852A.
Time Frame: Prior to Dose 1 and 6 Hours Post-Dose
Population: Only 9 patients had recorded values at 6 hours after treatment and were included in analysis.
Measure: Mean (95% Confidence Interval); unit: pg/mL
Groups:
- Patients Treated With 852A: Difference in range values from pre-treatment to post-treatment for cytokine level of TNF-a in patients treated with 852A.
Arm/Group | Patients Treated With 852A
Number analyzed (Participants) | 9
pg/mL | 8.26 [-10.10 to 26.63]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from beginning of study through 12 weeks (24 doses of study drug).
Description: Safety (toxicity) is one of the objectives of this study. Only serious adverse events were reported and collected as part of this study.
Arm/Group | Patients Treated With 852A Study Drug
Serious Adverse Events (participants affected / at risk) | 9/13
Other Adverse Events (participants affected / at risk) | 0/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Treated With 852A Study Drug (N=13)
Abdominal pain (Gastrointestinal disorders) | 1 (1) — Grade 3, severe
Acute idiopathic cardiomyopathy (Cardiac disorders) | 1 (1) — Grade 3, severe
Anorexia (Gastrointestinal disorders) | 1 (1) — Grade 3, severe
Cardiac left ventricular function (Cardiac disorders) | 1 (1) — Grade 2, moderate
Cardiac troponin levels increased (Cardiac disorders) | 1 (1) — Grade 4, life-threatening
Death due to Progressive Disease (General disorders) | 1 (1) — Grade 5, death
Dehydration (Gastrointestinal disorders) | 3 (3) — Grade 3, severe
Elevated liver enzymes (Hepatobiliary disorders) | 1 (1) — Grade 4, life-threatening
Fatigue (General disorders) | 1 (1) — Grade 3, severe
Gastrointestinal symptoms (Gastrointestinal disorders) | 1 (1) — Grade 3, severe
Infection/Febrile Neutropenia (Blood and lymphatic system disorders) | 3 (3) — Grade 3, severe
Nausea (Gastrointestinal disorders) | 1 (1) — Grade 3, severe
Pain (General disorders) | 3 (5) — Grade 3, severe
Renal failure (Renal and urinary disorders) | 1 (1) — Grade 3, severe
Renal, other (Renal and urinary disorders) | 1 (1) — Grade 3, severe
Vomiting (Gastrointestinal disorders) | 1 (1) — Grade 3, severe

LIMITATIONS AND CAVEATS:
Other Adverse Events that occurred were noted as targeted toxicities and not captured as adverse events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes